CLINICAL TRIAL: NCT01944150
Title: Interest of the Association of Two Complementary Techniques, Hypnosis and Transcutaneous Electrical Nerve Stimulation in the Treatment of Chronic Non-cancer Pain, Nociceptive and / or Neuropathic Pain: Randomized Trial
Brief Title: Association of Transcutaneous Electrical Nerve Stimulation and Hypnosis
Acronym: HYPTENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K121201; PHRI120049 (Other: Assistance Publique)
Record Dates: First submitted 2013-09-02; First posted 2013-09-17 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Limbs Arthrosis; Non Arthrosic Limbs Arthralgia; Chronic Lomboradiculalgia; Chronic Back Pain; Cervical Radiculopathy; Post-herpetic Neuralgia; Post-surgical Peripheral Neuropathic Pain; Post Trauma Neuropathic Pain; Complex Regional Pain Syndrome Type I or II; Tendinopathy
Keywords: Hypnosis; chronic pain; transcutaneous electrical nerve stimulation; nociceptive pain; neuropathic pain; complementary therapies
MeSH Terms: conditions — Radiculopathy; Neuralgia, Postherpetic; Complex Regional Pain Syndromes; Tendinopathy; Chronic Pain; Nociceptive Pain; Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation; Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS (Active Comparator): Patients with only transcutaneous electrical nerve stimulation (TENS),
  Interventions: Behavioral: Transcutaneous electrical nerve stimulation
- TENS and hypnosis. (Experimental): Patients with transcutaneous electrical nerve stimulation (TENS) and hypnosis simultaneously
  Interventions: Behavioral: Transcutaneous electrical nerve stimulation and hypnosis

INTERVENTIONS:
Behavioral: Transcutaneous electrical nerve stimulation — explanations about devices and their use are given to the patient during the first session. The right place where the electrodes should be placed on, the most effective programme (optimal electric frequency provided by the machine), intensity are tested by the nurse during 30 minutes lasting session
  Arms: TENS
Behavioral: Transcutaneous electrical nerve stimulation and hypnosis — explanations about devices and their use are given to the patient during the first session. The right place where the electrodes should be placed on, the most effective programme (optimal electric frequency provided by the machine), intensity are tested by the nurse. Following informations are collected by the second nurse: pain representation and its relief thoughts about a quiet place. TENS and hypnosis are associated in a unique 30 minutes session
  Arms: TENS and hypnosis.

SUMMARY:
At Saint-Antoine's hospital, in CETD a multidisciplinary team takes care of patients with chronic pain. Free-drug techniques are available to reduce their consumption of analgesics. This study is to assess the relief obtained by the simultaneous combination of these two techniques: transcutaneous electrical nerve stimulation and hypnosis.

DETAILED DESCRIPTION:
In the pain management centers, patients with chronic pain are supported by a multidisciplinary team. To optimize and reduce drug intake of analgesics, additional techniques (hypnosis, relaxation, cognitive behavioral therapy) and non-drug practices (transcutaneous electrical nerve stimulation) are offered to patients.

These techniques are most frequently performed by nurses and are used either separately or successively. The time interval during what the patient could expect pain relief is not known.

The hypothesis of the study is that simultaneous practice of two complementary therapies (transcutaneous electrical nerve stimulation (TENS) + hypnosis) decreases the intensity of pain in patients with chronic no cancer pain, nociceptive and/or neuropathic pain compared to practice of only one complementary therapy (TENS).

This study is an open randomized trial, comparative in two parallel groups (TENS versus TENS and hypnosis).

Trial design will be explained by the pain management center doctor. Inclusion and randomization performed by the nurse: group with TENS/group with TENS and hypnosis.

The patients will be followed up 8 times between day 0 and day180. Patients benefit from eight visits from day 0th to day 180th. Evaluations are EVA at each visit, SF36 questionnaires and score PGIC at one month, three and six months after the beginning of the strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 80 years suffering from chronic no cancer pain either nociceptive or neuropathic.
* The treated skin must not be wounded
* The patients must be able to comply with the requirement of the trial; they also need to express no objection to participate to this trial.
* Patient with social security

Exclusion Criteria:

* Patients with fibromyalgia, or having relaxation therapy sessions, acupuncture, cognitive and behavioral therapies
* Patients with cognitive disorders, an unaided hearing loss, a major hearing impairment, carrying a pace maker, having an allodynia or a complete anesthesia of the painful territory, a large spreader painful territory
* Sessions TENS practiced for analgesic by a professional within 3 years prior to inclusion, for the same pain (same features, same location)
* Renting at home a TENS device within 3 years prior to inclusion for analgesic
* Prior therapeutic care by hypnosis
* pregnant woman or having a desire of pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity | between the first visit and three months after the beginning of the strategy.
  The pain assessment is processed using a Visual Analog Scale (VAS), graduated from 0 to 100mm.
  The patient is asked to move a cursor on a line to reflect the severity of his/her pain. The left end indicates "no pain", the right one shows "the most intense pain you can imagine".
  On the other side, graduations are only seen by the caregiver. The pain intensity is read on this side, rated in millimetres.

SECONDARY OUTCOMES:
the patient's observance with the different strategies using a pad. | from one week after the beginning of the strategy up to 6 months.
  Collections of the data (number and duration of TENS device uses) from the patient log book
the consumption of analgesic | during 6 months.
  Collection of the concomitant treatments (processing) on the patient pad in every visit.
the quality of life estimated by the patient using the scale(ladder) SF36 and estimating the impression(printing) of change of the patient using the PGIC scale(ladder) | at the first visit, one month, three and six months after the beginning of the strategy, except the scale QDSA, which is used one, three and six months later after the beginning of the strategy.
  These two scales are self-assessment, exploring physical, emotional and social health.
  They allow pain impact assessment or professional activities, leisure activities and everyday life.
  The final aim is to identify if patients could recover their usual activity faster in one arm of the study versus the other one.

CONTACTS AND LOCATIONS:
Overall Officials: Louise GEOFFROY, Nurse, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CETD - Hospital Saint-Antoine, Paris, France

REFERENCES:
- [Derived] Smart KM, Ferraro MC, Wand BM, O'Connell NE. Physiotherapy for pain and disability in adults with complex regional pain syndrome (CRPS) types I and II. Cochrane Database Syst Rev. 2022 May 17;5(5):CD010853. doi: 10.1002/14651858.CD010853.pub3. PMID 35579382
- [Derived] Tonye-Geoffroy L, Mauboussin Carlos S, Tuffet S, Fromentin H, Berard L, Leblanc J, Laroche F. Efficacy of a combination of hypnosis and transcutaneous electrical nerve stimulation for chronic non-cancer pain: A randomized controlled trial. J Adv Nurs. 2021 Jun;77(6):2875-2886. doi: 10.1111/jan.14833. Epub 2021 Mar 30. PMID 33783846